CLINICAL TRIAL: NCT00896649
Title: Impact of Dedicated Breast Positron Emission Mammography vs. Conventional Two-View Digital Mammography on Recall Rates and Cancer Detection as a Screening Examination in Underserved Women
Brief Title: Positron Emission Mammography and Standard Mammography in Women at High Risk of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gustavo Mercier, BMC Attending Physician, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDR0000640404; BUMC-H-27136 (Other: BUMC IRB); W81XWH-06-1-0309 (Other: funding number); 05063002 (Other); HRPO #A-13777.2 (Other: DoD)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: PEM
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- positron emission mammography (Experimental): questionnaire administration digital mammography positron emission mammography
  Interventions: Other: questionnaire administration; Procedure: digital mammography; Procedure: positron emission mammography

INTERVENTIONS:
Other: questionnaire administration — Questionnaire regarding patient satisfaction with mammogram experience and with positron emission mammography experience.
Procedure: digital mammography — standard screening mammogram
Procedure: positron emission mammography — one-time positron emission mammography to compare recall rates with that of standard mammogram

SUMMARY:
RATIONALE: Screening tests may help doctors find cancer cells early and plan better treatment for breast cancer. It is not yet known whether positron emission mammography is more effective than standard mammography in finding breast tumors.

PURPOSE: This phase III trial is studying positron emission mammography to see how well it works compared with standard mammography in women undergoing screening mammogram at Boston Medical Center.

DETAILED DESCRIPTION:
OBJECTIVES:

* To install the breast Positron Emission Mammography system and to test and ensure its compliance with all regulatory agencies including the American College of Radiology and the Food and Drug Administration.
* To measure and compare the number of call-backs for positron emission mammography (PEM) imaging and conventional mammography.
* To measure and compare patient satisfaction for both conventional mammography and positron emission mammography in terms of comfort and pain.

OUTLINE: Patients undergo a conventional two-view mammogram and positron emission mammography (PEM). Immediately following treatment, patients complete a questionnaire on their satisfaction with the standard mammogram and the positron emission mammography.

After completion of study treatment, patients are followed annually.

ELIGIBILITY:
Inclusion criteria:

DISEASE CHARACTERISTICS:

* Scheduled to undergo screening mammogram at one of the Boston Medical Center-affiliated primary care clinics and meets 1 of the following criteria:

  * Dense breast tissue
  * At high-risk for breast cancer

PATIENT CHARACTERISTICS:

* Has 1 of the following racial or ethnic backgrounds based on the patient's country of birth or the mother and father's country of birth:

  * Hispanic
  * Haitian Creole
  * African American
  * Caucasian

PRIOR CONCURRENT THERAPY:

* None specified

Exclusion criteria:

* No history of breast cancer, palpable breast mass, abnormal nipple discharge, or other focal complaints warranting diagnostic mammogram

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2009-02; Primary Completion 2012-07 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Mercier, MD, PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Cancer Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not useful.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 193 participants were enrolled onto this study between 4/8/2009 through 5/31/2012 in the Breast Center.
Groups:
- Single Arm Positron Emission Mamm, Mammogram and Questionnaire: questionnaire administration positron emission mammography
  digital mammography: standard screening mammogram
  questionnaire administration: Questionnaire regarding patient satisfaction with mammogram experience and with positron emission mammography experience.
  positron emission mammography: one-time PEM to compare recall rates with that of standard mammogram
Period: Overall Study
Arm/Group | Single Arm Positron Emission Mamm, Mammogram and Questionnaire
Started | 193
Completed | 188
Not Completed | 5
Not completed — Physician Decision | 1
Not completed — Pregnancy | 1
Not completed — missing documentation | 1
Not completed — technical difficulties | 2

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Positron Emission Mammography (PEM), Mammography, Questionaire: questionnaire administration digital mammography positron emission mammography
  questionnaire administration: Questionnaire regarding patient satisfaction with mammogram experience and with positron emission mammography experience.
  digital mammography: standard screening mammogram
  positron emission mammography: one-time positron emission mammography to compare recall rates with that of standard mammogram
Arm/Group | Positron Emission Mammography (PEM), Mammography, Questionaire
Number analyzed (Participants) | 193
Age, Categorical [Count of Participants; unit: Participants] — Age of the subjects must be greater than or equal to 18 years of age.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 182
    >=65 years | 11
Sex/Gender, Customized [Count of Participants; unit: Participants] — The gender of the patient must be female per protocol.
  Participants
    Female | 193
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Hispanic/Non-Hispanic eligible
  Participants
    Hispanic or Latino | 8
    Not Hispanic or Latino | 185
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Caucasian African American
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 113
    White | 80
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Boston, Massachusetts, USA
  Participants
    United States | 193
Pregnancy status [Count of Participants; unit: Participants] — Only non-pregnant patients are allowed to participate.
  Participants
    negative pregnancy status | 192
    pregnant status | 1
No prior history of cancer in previous 5 years [Number; unit: participants] | 193

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Breast Imaging Assessment Reporting and Data System (BI-RADS) "0" Call-back in Mammography vs Breast Imaging Assessment Reporting and Data System (BI-RADS) "0" in Positron Emission Mammography
Description: Number of participants called back due to Breast Imaging Assessment Reporting and Data System (BI-RADS) "0" Mammogram compared to number of patients with Breast Imaging Assessment Reporting and Data System (BI-RADS) "0" in positron emission mammography
  Breast Imaging Assessment Reporting and Data System (BI-RADS) Scale:
  0 = Inconclusive for malignancy; call-back in mammography
  1. = normal
  2. = abnormal, with no malignancy
  3. = abnormal, likely benign
  4. = abnormal, likely malignant
  5. = malignant
Time Frame: immediately at completion of mammogram
Population: Number of participants who completed protocol with complete data set
Measure: Number; unit: participants
Groups:
- Single Arm Positron Emission Mammography and Questionnaire: questionnaire administration positron emission mammography
  digital mammography: standard screening mammogram
  questionnaire administration: Questionnaire regarding patient satisfaction with mammogram experience and with positron emission mammography experience.
  positron emission mammography: one-time positron emission mammography to compare recall rates with that of standard mammogram
Arm/Group | Single Arm Positron Emission Mammography and Questionnaire
Number analyzed (Participants) | 188
participants
  Number of BI-RAD "0" Mammogram | 28
  Number of BI-RAD "0" positron emission mammograph | 27

2. Secondary Outcome: Patient Satisfaction Level as Pertaining to Comfort and Pain for Each Study
Description: Number of participants satisfied with positron emission mammography with regard to comfort and pain for each study 1-7 rating scale, Entries from 1-4 considered Satisfied. Entries 5-7 considered not Satisfied.
Time Frame: One month
Population: All participants who completed imaging and questionnaires.
Measure: Number; unit: participants
Groups:
- Single Arm Positron Emission Mammo, Mammogram & Questionnaire: questionnaire administration positron emission mammography
  digital mammography: standard screening mammogram
  questionnaire administration: Questionnaire regarding patient satisfaction with mammogram experience and with PEM experience.
  positron emission mammography: one-time PEM to compare recall rates with that of standard mammogram
Arm/Group | Single Arm Positron Emission Mammo, Mammogram & Questionnaire
Number analyzed (Participants) | 188
participants
  Satisfied With Experience: Mammogram | 165
  Not Satisifed with Experience: Mammogram | 23
  Satisfied with the Experience: PEM | 175
  Not Satisfied with the Experience: PEM | 13

ADVERSE EVENTS:
Time Frame: There were no adverse events during the course of this study
Groups:
- Single Arm PEM, Mammography and Questionnaire: questionnaire administration positron emission mammography
  digital mammography: standard screening mammogram
  questionnaire administration: Questionnaire regarding patient satisfaction with mammogram experience and with PEM experience.
  positron emission mammography: one-time PEM to compare recall rates with that of standard mammogram
Arm/Group | Single Arm PEM, Mammography and Questionnaire
Serious Adverse Events (participants affected / at risk) | 0/188
Other Adverse Events (participants affected / at risk) | 0/188

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No